CLINICAL TRIAL: NCT03293706
Title: Evaluation of Carbohydrates (CHO): Tolerance, Breath Hydrogen and Methane
Brief Title: Evaluation of Carbohydrates Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BL37 Part 2
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Gastro-Intestinal Tolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CHO Control 1 Glucose (Active Comparator): 25 g glucose
  Interventions: Other: CHO Control 1 and 2 Glucose
- CHO Control 2 Glucose (Active Comparator): 25 g glucose
  Interventions: Other: CHO Control 1 and 2 Glucose
- CHO Experimental 1 Slowly Digested (Experimental): 25 g slowly-digested carbohydrate blend
  Interventions: Other: CHO Experimental 1 Slowly Digested
- CHO Experimental 2 Digestion Resistant (Experimental): 25 g digestion-resistant carbohydrate blend
  Interventions: Other: CHO Experimental 2 Digestion Resistant
- CHO Experimental 3 Low Sugar (Experimental): 25 g low sugar carbohydrate blend
  Interventions: Other: CHO Experimental 3 Low Sugar
- CHO Experimental 4 Maltodextrin (Experimental): 25 g maltodextrin
  Interventions: Other: CHO Experimental 4 Maltodextrin

INTERVENTIONS:
Other: CHO Control 1 and 2 Glucose — mixed in 237 ml/8 fl. oz. of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Control 1 Glucose; CHO Control 2 Glucose
Other: CHO Experimental 1 Slowly Digested — mixed in 237 ml/8 fl. oz. of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 1 Slowly Digested
Other: CHO Experimental 2 Digestion Resistant — mixed in 237 ml/8 fl. oz. of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 2 Digestion Resistant
Other: CHO Experimental 3 Low Sugar — mixed in 237 ml/8 fl. oz. of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 3 Low Sugar
Other: CHO Experimental 4 Maltodextrin — mixed in 237 ml/8 fl. oz. of a flavored non-caloric beverage; 1 time consumption
  Arms: CHO Experimental 4 Maltodextrin

SUMMARY:
The study is single-blind with a randomized, cross-over design to evaluate gastrointestinal tolerance of carbohydrate blends.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females in good health.
* Eligible to receive income in Canada and must demonstrate OHIP or equivalent medical coverage.

Exclusion Criteria:

* Subject with any type of food allergy or with a known history of AIDS, hepatitis, diabetes, cardio-vascular disease or GI disease.
* Subject taking medication, or with any condition which might, in the opinion of the PI either make participation dangerous to the subject or to others or affect the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Breath hydrogen | 0 to 7 hours
  Assessed in exhaled gasses

SECONDARY OUTCOMES:
GI tolerance symptoms | 0 to 48 hours
  Assessed using a subject tolerance questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided